CLINICAL TRIAL: NCT03683810
Title: The Effectiveness of Lactoferrin in the Management of Treatment-induced Anemia in Hematological Patients
Brief Title: The Effectiveness of Lactoferrin in the Management of Treatment-induced Anemia
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cyprus University of Technology (Other)
Collaborators: Hematological Clinic - Nicosia General Hospital (Unknown); German Oncology Center, Cyprus (Other); Limassol Hematology-oncology Center (Unknown)
Responsible Party: Principal Investigator, Dr. Andreas Charalambous, Associate Professor, Cyprus University of Technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AC-LFS-2018
Record Dates: First submitted 2018-09-24; First posted 2018-09-25 (Actual); Last update posted 2022-09-06 (Actual); Status verified 2022-09

CONDITIONS: Anemia
Keywords: hemoglobin; quality of life
MeSH Terms: conditions — Anemia | interventions — Lactoferrin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lactoferrin (Experimental): Participants will receive 4gr lactoferrin per day for a duration of 3 months + standard treatment for anemia
  Interventions: Dietary Supplement: Lactoferrin; Drug: Recombinant human erythropoietin
- Standard treatment (Active Comparator): Participants will receive only the standard treatment for anemia
  Interventions: Drug: Recombinant human erythropoietin

INTERVENTIONS:
Dietary Supplement: Lactoferrin — Lactoferrin in tablets 4g/daily
  Arms: Lactoferrin
Drug: Recombinant human erythropoietin — Recombinant human erythropoietin (rHuEPO, epoetin alfa)

SUMMARY:
This will be a randomised control trial designed to test the effectiveness of lactoferrin in the management of treatment-induced anemia in patients with hematological malignancies.

DETAILED DESCRIPTION:
Chemotherapy induced anemia (CIA) is a common adverse event in cancer patients reported to occur in 20-60% whilst the resulting low hemoglobin level is associated with impaired quality of life. Lactoferrin (LF) is a non-haem iron-binding protein that is part of the transferrin protein family, along with serum transferrin, ovotransferrin, melanotransferrin and the inhibitor of carbonic anhydrase, whose function is to transport iron in blood serum.

The aim of the study is to test the effectiveness of LF along with standard care in the management of treatment-induced anemia.

ELIGIBILITY:
Inclusion Criteria:

* Patients on active treatment (chemotherapy i.e. cyclophosphamide, doxorubicin, rituximab, cisplatin carboplatin, etoposide)
* Ability to independently complete the questionnaires

Exclusion Criteria:

* Allergy to Milk
* Lactose intolerance
* Celiac disease
* Patient of whom chemotherapy has been interrupted for more than 2 weeks (due to adverse effects)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-01-14 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin | Change from baseline at 2, 4, 6, 8, 10, 12
  Concentration of Hemoglobin levels in Serum

SECONDARY OUTCOMES:
Ferritin | Change from baseline at 2, 4, 6, 8, 10, 12
  Concentration of Ferritin Levels in Serum
Cytokine | Change from baseline at 2, 4, 6, 8, 10, 12 weeks
  Concentration of Cytokine Levels in Serum
LgG | Change from baseline at 2, 4, 6, 8, 10, 12 weeks
  Concentration of LgG Levels in Serum
LgA | Change from baseline at 2, 4, 6, 8, 10, 12 weeks
  Concentration of LgA Levels in Serum
LgM | Change from baseline at 2, 4, 6, 8, 10, 12 weeks
  Concentration of LgM Levels in Serum
General Quality of LIfe | Change from baseline at 4, 8, 12 weeks
  EQ-5d
Health related quality of life | Change from baseline at 4, 8, 12 weeks
  EORTC - QLQ C-30
Functional Assessment of Cancer Therapy Anemia | Change from baseline at 4, 8, 12 weeks
  FACT-An

CONTACTS AND LOCATIONS:
Overall Officials: Andreas CHARALAMBOUS, Principal Investigator — Cyprus University of Technology (Nursing Department)
Locations (2):
- Cyprus (2):
  - Hematology-Oncology Center, Limassol
  - Nicosia General Hospital, Nicosia

IPD SHARING:
Plan to Share IPD: No